CLINICAL TRIAL: NCT02865733
Title: Randomized Single-blind Study of Intravenous Maintenance of Remodulin® for the Treatment of Pulmonary Hypertension After Fontan Operation
Brief Title: Study of Remodulin® in Pediatric Pulmonary Hypertension With Single Ventricular Physiology After Fontan Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xu Zhuoming, chief cadiologist,Director of Cardiac intensive Care Unit, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SJTUMS-201607
Record Dates: First submitted 2016-08-01; First posted 2016-08-12 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Pulmonary Hypertension
Keywords: Remodulin®; pulmonary vascular resistance; univentricular physiology
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remodulin Injection (Experimental): Drug: Remodulin Injection Dosage:5 ng/kg/min-80ng/kg/min(0.15ml/hr-2.4ml/hr) Frequency: intravenous maintenance increase at a rate of 10ng/kg/min (0.3ml/hr)every 30 minutes Durations:48 hours
  Interventions: Drug: Remodulin
- Distilled water group (Placebo Comparator): Drug:distilled water Dosage:0.15ml/hr-2.4ml/hr Frequency:increase at a rate of 0.3ml/hr every 30 minutes Durations:48 hours
  Interventions: Drug: distilled water

INTERVENTIONS:
Drug: Remodulin — After Fontan operation, the mean pulmonary arterial pressure (mPAP)evaluated by CVP or transpulmonary pressure gradient(TPG) evaluated by Echo will be measured firstly, if the data met the criteria, and the patients were enrolled in the experimental group, the patients would be administrated intravenously of Remodulin® with the beginning of 5ng/kg/min, with the rate of 10ng/kg/min every 30 minutes up to 80ng/kg/min.
  Other Names: Treprostinil Injection
  Arms: Remodulin Injection
Drug: distilled water — After Fontan operation, the mPAP (evaluated by CVP) or TPG (evaluated by Echo) will be measured firstly, if the data met the criteria, and the patients were enrolled in placebo group, then the patients would be administrated intravenously of distilled water with the beginning of 0.15ml/hr, with the rate of 0.3ml/hr every 30 minutes up to 2.45ml/hr.
  Other Names: placebo
  Arms: Distilled water group

SUMMARY:
The aim of this study is to determine the safety and efficiency of Remodulin®（Treprostinil Injection）to reduce the pulmonary arterial pressure and prevent pulmonary hypertension (PH) after Fontan operation with univentricular physiology.

DETAILED DESCRIPTION:
PH is a significant contributor to the postoperative morbidity and mortality of congenital heart disease, especially after Fontan operation with univentricular physiology. Mild increase of pulmonary vascular resistance may lead to failure of Fontan circulation. Remodulin® has been approved for the treatment of adults with PH, but little is known about the effects in children with PH after Fontan operation. The study aim is to determine the safety and efficiency of Remodulin® to reduce the pulmonary arterial pressure and prevent PH in children after Fontan operation. Meanwhile pharmacokinetics of the drug were checked with or without the peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

After Fontan procedure, the criteria should be met

1. mPAP greater than 15 mmHg
2. TPG greater than 6 mmHg (exclude the obstruction of cavopulmonary anastomosis)

Exclusion Criteria:

After Fontan surgery :

1. Severe arrhythmia led to low cardiac output
2. Platelets smaller than 50,000*109/L and obvious bleeding

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
The primary end point is a composite variable | the first 48 hours after Remodulin used
  consisting of death, failing Fontan or failed Fontan according to high pulmonary vascular resistance

SECONDARY OUTCOMES:
Change from base line of pulmonary hemodynamic measurements | baseline and 48 hours
  Pp/Ps reduce >10% or TPG≤6mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuoming Xu, M.D.,Ph,D., Study Director — Cardiac intensive Care Unit,Department of Thoracic and Cardiovascular Surgery

REFERENCES:
- [Derived] Chen X, Cai XM, Zhang MJ, Xu JH, Li H, Xu ZM. Pharmacokinetics of treprostinil in children with functional single-ventricle pulmonary arterial hypertension: a randomized controlled trial. Ann Transl Med. 2021 Jul;9(14):1163. doi: 10.21037/atm-21-3188. PMID 34430604